CLINICAL TRIAL: NCT03121664
Title: A Phase 1, Open-label, Fixed-sequence Study To Estimate The Effects Of Multiple-dose Administration Of Itraconazole On The Steady-state Pharmacokinetics Of Pf-06649751 In Healthy Adult Subjects
Brief Title: A Study To Estimate The Effects Of Itraconazole On Pharmacokinetics Of Pf-06649751 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7601006; 2016-005201-39 (EudraCT Number)
Record Dates: First submitted 2017-04-07; First posted 2017-04-20 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Drug drug interaction, CYP3A4, itraconazole
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cohort 1 (Experimental)
  Interventions: Drug: PF06649751, Itraconazole

INTERVENTIONS:
Drug: PF06649751, Itraconazole — PF-06649751 0.25 mg on Days 1,2,3 PF-06649751 0.5 mg on Days 4,5,6 PF-06649751 1 mg on Days 7 to Day 25 Itracoanzole 200 mg on Days 12 to Day 25

SUMMARY:
The purpose of this study is to evaluate the impact of CYP3A4 inhibitor, itraconazole, on plasma concentration of PF-06649751 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

* Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.
* Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).

Unwilling or unable to comply with the Lifestyle Guidelines described in the protocol.

* Unwilling or unable to comply with the Lifestyle Requirements described in this protocol
* Subjects who had a history of allergy or intolerance to azole antifungal drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
PF-06649751 and PF-06752844 steady state Cmax | Day 11 and Day 25
  Maximum Observed Plasma Concentration
PF-06649751 and PF-06752844 steady state AUC24 | Days 11 and Day 25
  Area Under the Curve From Time Zero to the end of the dosing period

SECONDARY OUTCOMES:
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Day 0
  C-SSRS assess whether participant experience the following: completed suicide (1), suicide attempt (2) (response "YES" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("yes" on "preparatory acts or behavior"), suicidal ideation (4) ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific pan and intent), any suicidal behavior or ideation, self-injurious behavior (7) ("yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Day 7
  C-SSRS assess whether participant experience the following: completed suicide (1), suicide attempt (2) (response "YES" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("yes" on "preparatory acts or behavior"), suicidal ideation (4) ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific pan and intent), any suicidal behavior or ideation, self-injurious behavior (7) ("yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Day 14
  C-SSRS assess whether participant experience the following: completed suicide (1), suicide attempt (2) (response "YES" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("yes" on "preparatory acts or behavior"), suicidal ideation (4) ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific pan and intent), any suicidal behavior or ideation, self-injurious behavior (7) ("yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Day 21
  C-SSRS assess whether participant experience the following: completed suicide (1), suicide attempt (2) (response "YES" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("yes" on "preparatory acts or behavior"), suicidal ideation (4) ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific pan and intent), any suicidal behavior or ideation, self-injurious behavior (7) ("yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Day 26
  C-SSRS assess whether participant experience the following: completed suicide (1), suicide attempt (2) (response "YES" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("yes" on "preparatory acts or behavior"), suicidal ideation (4) ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific pan and intent), any suicidal behavior or ideation, self-injurious behavior (7) ("yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Day 1 to Day 26
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Y days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug X was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601006&StudyName=A+Phase+1%2C+Open-label%2C+Fixed-sequence+Study+To+Estimate+The+Effects+Of+Multiple-dose+Administration+Of+Itraconazole+On+The+Steady-state+Pharmacokinetics+Of+Pf-06649751+In+Healthy+Adult+Subjects